CLINICAL TRIAL: NCT04600817
Title: A Phase 2, Randomized, Single-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of TJ107 in Lympopenic Patients With Newly Diagnosed Glioblastoma Who Completed Standard Concurrent Chemoradiotherapy (CCRT)
Brief Title: A Study to Evaluate the Efficacy and Safety of TJ107 in Lympopenic Patients With Newly Diagnosed Glioblastoma Who Completed Standard Concurrent Chemoradiotherapy (CCRT)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TJ Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJ107001GBM201
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Newly Diagnosed Glioblastoma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TJ107 (Experimental)
  Interventions: Drug: TJ107
- TJ107Placebo (Placebo Comparator)
  Interventions: Drug: TJ107 placebo

INTERVENTIONS:
Drug: TJ107 — QW8
  Arms: TJ107
Drug: TJ107 placebo — QW8
  Arms: TJ107Placebo

SUMMARY:
A Phase 2, Randomized, Single-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of TJ107 in Lympopenic Patients with Newly Diagnosed Glioblastoma Who Completed Standard Concurrent Chemoradiotherapy (CCRT)

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF)
2. Age ≥ 18 years and ≤70 years.
3. Gross total resection equal to or greater than 80% based on post-op MRI, compared to pre-op MRI (Patients requiring biopsy only is not eligible)
4. Patients newly diagnosed with glioblastoma either radiologically or pathologically and completed concurrent chemo-radiotherapy (CCRT) with plan to receive adjuvant temozolomide therapy with curative intent
5. Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to the randomization.1) Absolute lymphocyte count (ALC) ≤1×109/L. 2) Absolute neutrophil count (ANC) ≥ 1.5×109/L. 3) Platelet count ≥ 100×109/L (without transfusion within 14 days prior to Cycle 1, Day 1). 4) Hemoglobin ≥ 9 g/dL Patients may be transfused or may receive erythropoietic treatment as per local standard of care. 5) Total bilirubin ≤ 1.5 × the upper limit of normal (ULN). 6) AST and ALT ≤ 3 × ULN. 7) Alkaline phosphatase ≤ 2.5 × ULN (For subject with proven liver or bone metastasis, alkaline phosphatase ≤ 5 × ULN is allowed). 8) Serum albumin ≥ 2.5 g/dL. 9) Serum creatinine ≤ 1.5 mg/dL. 10) Prothrombin time (PT) and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN. This applies only to patients who are not receiving therapeutic anticoagulation. Patients receiving therapeutic anticoagulation should be on a stable dose
6. Karnofsky score ≥ 60
7. Life expectancy > 12 weeks
8. For women of childbearing potential*: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year from the date of informed consent to at least 3 months after the last dose of study drugs. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below: With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 3 months after the last dose of study treatment (TJ107) and 6 months after the last dose of temozolomide to avoid exposing the embryo. Men must refrain from donating sperm during this same period. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence and withdrawal are not acceptable methods of contraception.

   * A woman is of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
   * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, and established proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
   * Hormonal contraceptive methods must be supplemented by a barrier method plus spermicide.
   * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception

Exclusion Criteria:

1. Subjects receiving 21 days hypofractionated radiotherapy due to clinical condition
2. Multifocal glioma (≥3 lesions)
3. Patients with primary subtentorial glioblastoma multiforme
4. Patients who have evidence of leptomeningeal disease
5. Patients on corticosteroid treatment have not a stable or decreasing dose for 14 days before randomization.
6. Pregnancy, lactation, or breastfeeding (with lactation or breastfeeding required during the study period)

   *Serum pregnancy test for women of childbearing potential (including women who have had a tubal ligation) must be performed and documented as negative within 14 days prior to randomization
7. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 3 months, unstable arrhythmias, and/or unstable angina
8. Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, and inherited liver disease or current alcohol abuse
9. Poorly controlled Type 2 diabetes mellitus defined as a screening hemoglobin A1C ≥ 8% or a fasting plasma glucose ≥ 160 mg/dL (or 8.8 mmol/L)
10. Anticipation of need for a major surgical procedure (requiring general anesthesia) during the study period
11. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension (defined by blood pressure higher than 150/90mmHg despite effective anti-hypertensive treatments) and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in trial or which would jeopardize compliance with the protocol
12. Any anti-cancer therapy, whether investigational or approved, including chemotherapy, immunotherapy, gene therapy, cancer vaccine, cell therapy, cytokines, hormonal therapy, and/or radiotherapy) received after standard concurrent chemo-radiotherapy (CCRT)
13. Persisting toxicity related to prior therapy (NCI CTCAE v. 5.0 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable
14. Malignancies other than disease under study within 5 years prior to randomization except for those with a negligible risk of metastasis or death (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, or ductal carcinoma in situ)
15. Uncontrolled hypercalcemia (ionized Calcium > 1.5 mmol/L or Calcium > 12 mg/dL or adjusted serum Calcium ≥ ULN) or symptomatic hypercalcemia requiring bisphosphate or denosumab

    *Patients without history of clinically significant hypercalcemia, receiving either bisphosphonate or denosumab prophylactically is eligible

    ** Denosumab receiving patients should agree to switch to bisphosphate, and not contraindicated for bisphosphate use are eligible
16. Patients with active virus infection requiring systemic treatment at screening 1) Positive test for HIV infection 2) Active HBV hepatitis: positive for HBsAg and HBV-DNA, if HBsAg positive but HBV-DNA negative during the screening can participate in the study.3) Active HCV hepatitis: positive for hepatitis C virus (HCV) antibody and HCV RNA. But the subject can be enrolled with serum anti-HCV positive and HCV RNA negative.
17. Patients with autoimmune disease requiring treatment at the time of screening (appendix 3. List of autoimmune disease)1) Patients with adrenal or pituitary insufficiency requiring physiological dose of corticosteroid such as tyrosine, insulin. 2) Patients with leukoplakia, resolved pediatric asthma, atopic dermatitis, type 1 diabetic, hypothyroidism due to autoimmune disease only requiring hormone replacement therapy, psoriasis not requiring systemic treatment, and other disease status that recurrence nor exacerbations are not expected unless there is external contributing factors
18. Administration of a live, attenuated vaccine within 14 days before randomization or anticipation that such a live attenuated vaccine will be required during the study.1) Measles, mumps, rubella, chickenpox, yellow fever, rabies, Bacillus Calmette-Guérin, BCG, herpes zoster, typhoid vaccines. 2) Seasonal influenza vaccine in injection formulation are generally not live vaccine, thus are allowed. Yet intra-nasal influenza vaccine such as Flumist® is attenuated live vaccine, thus is not allowed
19. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
20. Severe infections within 2 weeks prior to randomization, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
21. Prior allogeneic bone marrow transplantation or prior solid organ transplantation
22. Treatment with systemic immunosuppressive medications (including daily prednisone > 30mg, dexamethasone > 5mg, or equivalent dose of corticosteroid, cyclophosphamide, azathioprine, methotrexate, thalidomide, and TNF-α antagonists but not limited to) within 2 weeks prior to randomization. 1) Patients who acutely receives low dose immunosuppressive medication (e.g. daily prednisone ≤ 30 mg or daily dexamethasone ≤ 5 mg) can be enrolled upon approval from study medical monitor. 2) The use of inhaled corticosteroids (e.g., fluticasone for chronic obstructive pulmonary disease) is allowed. 3) The use of oral mineralocorticoids (e.g., fludrocortisone for patients with orthostatic hypotension) is allowed.
23. History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis * History of radiation pneumonitis in the radiation field (fibrosis) is allowed."

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-12-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with average of ALC at 3w after first TJ107 dose and at pre-dose 3rd TMZ ≥1.5X109/L | 18 months

CONTACTS AND LOCATIONS:
Locations (16):
- China (15):
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Tangdu Hospital of The Fourth Military Medical University of Chinese PLA, Xi'an, Shaanxi
  - Beijing Tiantan Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Chongqiong Cancer Hospital, Chongqing
  - Huashan Hospital Affiliated to Fudan University, Shanghai
  - Tianjin Huanhu Hospital, Tianjin
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided